CLINICAL TRIAL: NCT01017250
Title: Radiosurgery and Avastin for Recurrent Malignant Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018943
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Malignant Glioma
Keywords: Recurrent
MeSH Terms: conditions — Glioma; Recurrence | interventions — Radiosurgery; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental): Avastin and Radiosurgery
  Interventions: Radiation: Stereotactic Radiosurgery (SRS); Drug: Bevacizumab

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (SRS) — Tumor Volume < 2.0cm receives 24 Gy in 1 fraction Tumor Volume 2.0-2.9cm receives 18 Gy in 1 faction Tumor Volume 3.0-4.9cm receives 25 Gy in 5Gy/fraction
Drug: Bevacizumab — Bevacizumab (Avastin) 10 mg/kg given the day before SRS and 2 weeks after SRS
  Other Names: Avastin

SUMMARY:
The purpose of this study is to assess the central nervous system (CNS) toxicity in patients with recurrent malignant gliomas treated with concurrent Avastin and stereotactic radiosurgery (SRS).

DETAILED DESCRIPTION:
In this pilot study, 15 human subjects with recurrent, unifocal malignant gliomas up to 5-cm in maximum dimension no longer responding to conventional chemotherapy but able to tolerate further chemotherapy will be enrolled. The primary endpoint of this study will be the proportion of patients who experience CNS toxicity, with secondary endpoints progression-free survival, overall survival, steroid dosage, development of radionecrosis, quality of life, objective radiographic response and performance status.

ELIGIBILITY:
Inclusion Criteria:

* History of malignant glioma (WHO Grade III or IV) of the brain treated with some combination of surgery, biochemotherapy and conventionally fractionated external beam radiotherapy
* Radiotherapy completed at least 6 months prior to recurrence
* Age 18 years and older
* New or enlarging contrast-enhancing and/or 18FDG-avid nodule, at least 1 cm diameter
* Estimated life expectancy of 3 months or longer

Exclusion Criteria:

* Avastin therapy within 21 days of start of participation
* Contraindication to Avastin therapy or brain MRI
* Presence of bleeding diathesis or coagulopathy
* History of prior arterial thrombotic event, myocardial infarction, angina, CVA, TIA, CABG angioplasty or stenting within 6 months.
* Inadequately controlled hypertension (defined as systolic blood pressure
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Clinically significant vascular disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to onset of treatment
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of abdominal fistula or GI perforation within 6 months prior to onset of treatment
* Serious non-healing wound, active ulcer or untreated bone fracture
* Proteinuria demonstrated by Urine Protein Creatinine ratio > 1.0
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkpatrick, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Radiation Oncology, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period Jan 2, 2010-Jan 12, 2011 Location: Radiation Oncology Clinic
Groups:
- Stereotactic Radiosurgery: Avastin 10 mg/kg given intravenously (IV) within 24 hours before and two weeks following their first treatment with Stereotactic Radiosurgery (SRS).
  SRS is
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery
Started | 15
2-month MRI | 14 (1 participant did not return for the 2 month MRI at treating facility. Resides out of state.)
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.27 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Toxicity
Description: Number of participants who experience Grade 3 or higher adverse events in the "Nervous System Disorder" domain of Common Toxicity Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: 2 months after Stereotactic Radiosurgery
Population: The number of participants with CNS toxicity is reported.
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
participants | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in months from the start of stereotactic radiosurgery (SRS) to the date of first progression according to Revised Assessment in Neuro-Oncology (RANO)criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve. Per RANO, progression is defined as a 20% increase in the sum of the longest diameter of target lesions,or a measurable increase in a non-target lesion or the appearance of new lesions.
Time Frame: 1 year
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
months | 3.9 [2.0 to 5.1]

3. Secondary Outcome: Radiographic Response at Month 2
Description: Radiographic response at 2 months after stereotactic radiosurgery (SRS) assessed by MRI and based on modified Response Assessment in Neuro-Oncology (RANO) criteria.Per RANO, complete response (CR) is the disappearance of all target lesions;Partial Response(PR)is a >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 2 months after SRS
Population: Intent to treat
Measure: Number; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
Participants
  Complete response | 0
  Partial Response | 0
  Stable Disease | 10
  Progressive Disease | 4
  Not Evaluable | 1

4. Secondary Outcome: Overall Survival(OS)
Description: Time in months from the start of stereotactic radiosurgery (SRS) to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 2 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
months | 14.4 [6.0 to 18.3]

5. Secondary Outcome: Change in Quality of Life From Baseline to 2 Months After Stereotactic Radiosurgery (SRS)
Description: Quality of life as measured by the change in Functional Assessment of Cancer Therapy-Brain (FACT-Br) scores from baseline to 2 months after SRS. The FACT-Br (version 4) is comprised of the Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item core questionnaire evaluating the domains of physical, family/social, emotional and functional well-being, with the addition of 23 brain cancer specific questions. The FACT-G total score is the sum of the four FACT-G domain scores. The Brain Cancer Subscale (BrCS) is the sum of 19 brain cancer specific questions. The FACT-Br Trial Outcome Index (TOI) is the sum of the BrCS score and the physical and family/social domain scores. The FACT-Br total score is the sum of the FACT-G total score and the BrCS score. Higher scores for all scales indicate improved quality of life (QOL).Change score = score at 2 months after SRS - score at baseline. Positive change scores indicate improved quality of life.
Time Frame: 2 months after SRS
Population: Intent to Treat; only 10 patients out of 15 completed the month 2 questionnaire.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 10
units on a scale
  FACT-G: physical well-being ( range: 0-28) | -2.9 (1.0)
  FACT-G: Family/Social Well-being ( range: 0-28) | -0.1 (0.9)
  FACT-G: Emotional Well-being ( range: 0-24) | -0.4 (1.4)
  FACT-G: Functional Well-being ( range: 0-28) | -1.2 (1.3)
  FACT-G: Total Score ( range: 0-108) | -4.6 (3.8)
  FACT-Br: BrCS ( range: 0-76) | 0.8 (2.7)
  FACT-Br: TOI ( range: 0-132) | -3.2 (3.6)
  FACT-Br: Total Score ( range: 0-184) | -3.7 (4.9)

6. Secondary Outcome: Cognition at 2 Months After Stereotactic Radiosurgery (SRS)as Measured by the Mini-Mental State Exam ( MMSE)
Description: Cognition as measured by the change in the Mini-Mental State Exam (MMSE) scores from baseline to 2 months after SRS. The MMSE is an 11-item measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall and language. The maximum score is 30. Change score = score at 2 months after SRS - score at baseline. Higher scores for this scale indicate improved quality of life(QOL). Positive change scores indicate improved cognition.
Time Frame: 2 months after SRS
Population: Intent to Treat: only 14 patients out of 15 completed the month 2 questionnaire
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 14
units on a scale | 0.3 (0.2)

7. Secondary Outcome: Cognition at 2 Months After Stereotactic Radiosurgery (SRS) as Measured by the Trail Making Test (TMT)
Description: Cognition as measured by the change in scores on the Trail Making Test (TMT). The TMT consists of two parts. Part A (TMT-A) requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for Part B (TMT-B) except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task. Shorter time scores indicates improved cognition. Change score = score at 2 months after SRS - score at baseline. Negative change scores indicate improved cognition.
Time Frame: 2 months after SRS
Population: Intent to treat: only 14 of 15 patients completed the month 2 questionnaire
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 14
seconds
  TMT-A | 0.6 (3.3)
  TMT-B | -15.5 (9.4)

8. Secondary Outcome: Performance Status at 2 Months After Stereotactic Radiosurgery (SRS)
Description: Number of patients with a 10% decline in Karnofsky Performance Status (KPS) from baseline to 2 months after SRS. KPS is rated on a 0 to 100 scale representing a patient's ability to perform normal activity, ability to do active work, and the need for assistance. A score of 100 is "perfect" health and 0 represents death.
Time Frame: 2 months after SRS
Population: Intent to Treat: only 13 out of 15 patients completed month 2 KPS scores
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 13
participants | 11

9. Secondary Outcome: Steroid Usage After Stereotactic Radiosurgery (SRS)
Description: Number of patients using steroids at baseline and at 2 months after SRS.
Time Frame: 2 months after SRS 2 months after SRS 2 months after SRS
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 15
participants
  Baseline | 2
  2 months after SRS | 4

10. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 1 Week After Stereotactic Radiosurgery (SRS): K-trans
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. K-trans is the widely accepted MR method for quantitating brain tumor microvascular permeability( a measure of blood transport.) K-trans will indicate a combination of both flow and permeability properties of tissue. K-trans will indicate the tissue perfusion per unit volume, with a reduction in K-trans suggesting an increased anti-tumor effect and potentially improved outcome. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 1 week after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-2) min(-1)
Groups:
- Stereotactic Radiosurgery: Avastin 10 mg/kg given intravenously (IV) within 24 hours before and two weeks following their first treatment with Stereotactic Radiosurgery (SRS).
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-2) min(-1)
  Baseline | 6.7 [0.6 to 11.0]
  One week post SRS | 4.1 [0.0 to 6.0]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.04, Wilcoxon signed rank

11. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 2 Months After Stereotactic Radiosurgery (SRS): K-trans
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. K-trans is the widely accepted MR method for quantitating brain tumor microvascular permeability( a measure of blood transport.) K-trans will indicate a combination of both flow and permeability properties of tissue. K-trans will indicate the tissue perfusion per unit volume with a reduction in K-trans suggesting an increased anti-tumor effect and potentially improved outcome. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 2 months after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-2) min(-1)
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-2) min(-1)
  Baseline | 6.7 [0.6 to 11.0]
  2 months after SRS | 0 [0 to 0.0]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.002, Wilcoxon signed rank

12. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 1 Week After Stereotactic Radiosurgery (SRS): AUC
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. Area under the curve (AUC) is utilized to measure the signal enhancement ratio washout volume and could be predictive of cancer treatment response. It is possible AUC could be used as a prognostic indicator of the eventual response. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 1 week after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: mmol/kg∙s
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
mmol/kg∙s
  Baseline | 2.1 [1.0 to 2.7]
  One week post SRS | 1.4 [0.5 to 2.1]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank

13. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 2 Months After Stereotactic Radiosurgery (SRS): AUC
Description: as for outcome 12
Time Frame: 2 months after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: mmol/kg∙s
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
mmol/kg∙s
  Baseline | 2.1 [1.0 to 2.7]
  2 months after SRS | 0.1 [0.0 to 0.5]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.0005, Wilcoxon signed rank

14. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 1 Week After Stereotactic Radiosurgery (SRS): EVF
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. By measuring extracellular extravascular volume fraction (EVF) it is possible to gain information on brain tissue perfusion. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 1 week after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-1)
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-1)
  Baseline | 0.58 [0.1 to 1.1]
  One week post SRS | 0.48 [0.0 to 0.9]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.53, Wilcoxon signed rank

15. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 2 Months After Stereotactic Radiosurgery (SRS): EVF
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 2 months after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-1)
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-1)
  Baseline | 0.58 [0.1 to 1.1]
  2 months after SRS | 0 [0 to 0.0]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.002, Wilcoxon signed rank

16. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 1 Week After Stereotactic Radiosurgery (SRS): ADC
Description: DCE-MRI is a quantitative method that allows for non-invasive analysis of tumor vascular characteristics. Diffusion-weighted imaging, dependent on motion of water molecules, provides information regarding tissue integrity. Apparent diffusion coefficient (ADC) values in the normal brain parenchyma, and those in brain tumors were measured. Patients had a DCE-MRI at baseline and at 1 week and 2 months after SRS.
Time Frame: 1 week after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-6) mm^2/s
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-6) mm^2/s
  Baseline | 980 [830 to 1130]
  One week post SRS | 980 [830 to 1080]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.76, Wilcoxon signed rank

17. Secondary Outcome: Dynamic Contrasted-enhanced MRI (DCE-MRI) Perfusion Indices at 2 Months After Stereotactic Radiosurgery (SRS): ADC
Description: as for outcome 16
Time Frame: 2 months after SRS
Population: Intent-to-treat; only 12 of 15 patients had DCE-MRI results at both time points.
Measure: Median (Inter-Quartile Range); unit: 10(-6) mm^2/s
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 12
10(-6) mm^2/s
  Baseline | 980 [830 to 1130]
  2 months after SRS | 990 [830 to 1240]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; This was a test on the change from baseline to the post-SRS time point for all patients; Test type: Superiority or Other; p = 0.34, Wilcoxon signed rank

ADVERSE EVENTS:
Arm/Group | Stereotactic Radiosurgery
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery (N=15)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Radiosurgery (N=15)
Tinnitus (Ear and labyrinth disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 6
Gait disturbance (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 3
Confusion (Psychiatric disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No